CLINICAL TRIAL: NCT06492746
Title: Assessing for Personalized Blood Pressure Targets During Cardiopulmonary Bypass With the Proprietary Cerebral Adaptive Index: A Pilot Investigation
Brief Title: Personal BP - CAI Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-15
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cardiopulmonary bypass patients receiving blood pressure and oximetry monitoring (Experimental)
  Interventions: Device: HemoSphere Advanced Monitoring Platform with Acumen IQ sensor and Tissue Oximetry Monitoring

INTERVENTIONS:
Device: HemoSphere Advanced Monitoring Platform with Acumen IQ sensor and Tissue Oximetry Monitoring — The arterial line with Acumen IQ sensor and Foresight Elite sensor will be connected to the HemoSphere monitor with laptop displaying the CAI parameter.

SUMMARY:
A single-center, prospective, observational pilot of the Cerebral Adaptive Index for assessing personalized blood pressure targets

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 45 years
3. Planned cardiac surgery with Cardiopulmonary Bypass (CPB)
4. Planned monitoring with ForeSight sensor and HemoSphere monitor
5. Planned arterial catheterization for blood pressure monitoring
6. High risk for cerebral vascular disease, defined as: a history of hypertension, pulse pressure > 60 mmHg, diabetes, stroke, transient ischemic attack, carotid bruit, tobacco smoking, or peripheral vascular disease

Exclusion Criteria:

1. Non-English speaking
2. Confirmed to be pregnant
3. Surgery for congenital heart defect
4. Non-availability of HemoSphere with laptop CAI interface

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To determine the magnitude and duration of CAI | Duration of the procedure through 30 days
  To determine the sum of the product of magnitude and duration that CAI during cardiopulmonary bypass (CPB) is at or above the threshold of 45 during current standard of care and assess the incidence of CAI ≥45 in the absence of decreased cerebral StO2 or MAP thresholds.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Hospital, Evanston, Illinois, United States